CLINICAL TRIAL: NCT00843323
Title: Histological and Immunohistochemical Study of Photodamaged Skin Submitted to MAL-PDT
Brief Title: Photodynamic Therapy (PDT) Effect on Large Surface Photodamaged Skin
Acronym: PDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Regensburg (Other)
Responsible Party: Principal Investigator, Luis Antonio Torezan, ASSOCIATE PROFESSOR OF DERMATOLOGY, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0614/08
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Actinic Keratosis; Photoaging; Solar Elastosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Methylaminolevulinate - photodynamic therapy — Methylaminolevulinate cream 16% applied for 3 hours under occlusion on the face and then illuminated with red LED device

SUMMARY:
In this study, 26 patients were selected and included for full-face photodynamic therapy sessions. All patients presented signs of photoaging skin and multiple actinic keratosis. Photographs and Biopsies were taken before and after the procedure. Clinical and histological aspects as well as immunohistochemical aspects regarding neocollagen induction and tumor expression were evaluated.

DETAILED DESCRIPTION:
Study design:

Patients and methods:

26 patients (16 females, 8 males) age 35-90 years, mean 59,4 y Skin types I-IV, severely photodamaged facial skin Multiples Aks on the face ( total 268) minimum of 3 per patient Approved by local ethical committee and informed consent given

Treatment procedure:

Prior curettage Full-face MAL application ( Metvix ®, Galderma France) 1,5 tube per treatment Incubation time 3 hs - in the first treatment session; and 1,5 h - in the 2 nd and 3 rd sessions Illumination LED (Aktilite® Photocure, Norway) 635 nm 37 J/cm2 3 treatments performed, one month apart Pain monitoring: forced air cooling device

Evaluation:

Clinical - 5 point scale based on Dover's and Zane's studies Dover JS et al. Topical ALA combined with IPL in photoaging. Arch Dermatol 2005; 141: 1247-52 Zane et al. Clinical and echographical analysis of MAL- PDT in photodamaged skin. Laser Surg Med 2007; 39: 203-9

Histological - Hematoxilin- Eosin staining

Immunohistochemical study- HP 53, Metalloproteinases, Procollagen I,

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe photodamage and at least 3 actinic keratosis on the face

Exclusion Criteria:

* Pregnancy, laser, chemical peel, imiquimod or 5-Fu treatment in the last year

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Torezan, MD, Principal Investigator — Hospital das Clinicas - Faculdade de Medicina USP - Sao Paulo- Brazil